CLINICAL TRIAL: NCT00271336
Title: Pentoxifylline in the Treatment of Necrotizing Enterocolitis in Premature Neonates
Brief Title: Pentoxifylline in the Treatment of NEC in Premature Neonates
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Cathy Hammerman, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: chammerman1
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2005-12

CONDITIONS: Necrotizing Enterocolitis
Keywords: NEC; Premature Infants; TNF; Pentoxifylline
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator)
  Interventions: Drug: Pentoxifylline
- B (Experimental)
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pentoxifylline

SUMMARY:
Pentoxifylline improves microcirculation and decreases TNF alpha levels associated with sepsis, rendering it of potential therapeutic value in necrotizing enterocolitis in premature neonates.

DETAILED DESCRIPTION:
Preterm neonates with a clinical suspicion of necrotizing enterocolitis (NEC) will potentially be candidates for study. After obtaining parental consent, the infants will be prospectively and randomly assigned to one of two groups: 1. Treatment group: to receive IV pentoxifylline (5 mg/kg/hour to run over 6 hour x 6 days) and 2. Placebo group: to receive an equal volume of ½ normal saline to run over 6 hours x 6 days.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants <1750 gm. birth weight
* Abdominal x-ray consistent with NEC (dilated loops, bowel wall edema, fixed or persistent dilated loop with (or without pneumatosis)

Exclusion Criteria:

* Abdominal perforation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that fewer of the babies who are treated with PTX will progress to serious NEC related morbidity, ie. perforation, surgery [including peritoneal drain placement], and/or death related to NEC. | Three years

SECONDARY OUTCOMES:
To demonstrate lower levels of TNF alpha,fecal calprotectin;Improved SMA blood flow;Quicker radiographic resolution; Decreased feeding intolerance after acute NEC episode; and lower NEC associated long term morbidity. | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Hammerman, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel